CLINICAL TRIAL: NCT02601638
Title: Effect of Total Laryngectomy Preoperative Education on Postoperative Complications and Unplanned Hospital Readmission
Brief Title: Laryngectomy Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201411097
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Total Laryngectomy
MeSH Terms: interventions — Demography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): * Demographics and Health History Questionnaire (5-10 minutes to complete)
  * Pre-Class Laryngectomy Survey (5-10 minutes to complete)
  * Attend a preoperative counseling session with a speech pathologist. It will take 30-60 minutes
  * Attend the Total Laryngectomy Preoperative Education Class. Participants will attend within 1-2 weeks of providing written consent and prior to their scheduled surgery. The preoperative education class will take one hour.
  * Complete the Day of Hospital Discharge Laryngectomy Survey at the time of discharge from the hospital (5-10 minutes to complete)
  * Perform the day of discharge practicum assessing the minimal competency skills for laryngectomy care prior to discharge from the hospital.
  * Complete the Laryngectomy Education Study Exit survey. Participants will perform an exit survey at the first clinic appointment after 30 days after hospital discharge (15-30 minutes to complete)
  Interventions: Other: Demographics and Health History Questionnaire; Other: Pre-Class Laryngectomy Survey; Behavioral: Counseling session with speech pathologist; Behavioral: Total Laryngectomy Preoperative Education Class; Other: Day of Hospital Discharge Laryngectomy Survey; Other: Day of Discharge Practicum; Other: Laryngectomy Education Study Exit Survey

INTERVENTIONS:
Other: Demographics and Health History Questionnaire
Other: Pre-Class Laryngectomy Survey
Behavioral: Counseling session with speech pathologist
Behavioral: Total Laryngectomy Preoperative Education Class
Other: Day of Hospital Discharge Laryngectomy Survey
Other: Day of Discharge Practicum
Other: Laryngectomy Education Study Exit Survey

SUMMARY:
Patients undergoing total laryngectomy are at high risk for 30-day unplanned readmission. Many of these readmissions are related to stomal care, and it is thought that the readmissions could be prevented with better patient and caregiver education. The investigators are studying the effect of a comprehensive perioperative education program on 30-day unplanned readmission for patients undergoing total laryngectomy.

The comprehensive perioperative education program will include the following additional interventions:

-Preoperative visit with the speech pathologist for explanation of laryngectomy physiology, stomal education, and alaryngeal voice rehabilitation. Participants will be expected to undergo this intervention and to attend it with their "laryngectomy coach" (a family member or friend to accompany the patient through the education process), but failure to meet with the speech pathologist will not exclude a patient from the study.

* Preoperative education class with a designated ENT laryngectomy nurse for patient and caregiver. The hands-on class introduces the patient and laryngectomy coach to the basics of stomal care. Participants and their "laryngectomy coach" will be expected to attend the preoperative education class
* Printed laryngectomy journey guide given to patients at time of study enrollment for patient/caregiver. This journey guide details the preoperative, in-hospital, and post-discharge course and is provided as a reference throughout their journey.
* Formalized, nursing administered practical evaluation of minimal competency of laryngectomy care for patient and caregiver/laryngectomy coach.

This study will follow patients prospectively from the time of study commencement and then assess changes in patient knowledge before and after the education intervention. It will also compare rate of stomal complications and readmission rates to institutional historical averages to assess improvement in quality care.

ELIGIBILITY:
Inclusion Criteria:

* planned total laryngectomy at Barnes Jewish Hospital
* age 18 or older
* understand spoken or written English language
* able to provide informed consent.

Exclusion Criteria:

-none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Rate of 30-day unplanned readmission | 30 days after hospital discharge (approximately 7 weeks after registration)
  -Calculate and report the rates of readmission for the patients undergoing the comprehensive laryngectomy education and compare to the rates of unplanned readmission and postoperative complications from historical cohorts at our institution.
Rate of postoperative complications | 30 days after hospital discharge (approximately 7 weeks after registration)
  -Calculate and report the rates of readmission for the patients undergoing the comprehensive laryngectomy education and compare to the rates of unplanned readmission and postoperative complications from historical cohorts at our institution.
Change in patient's knowledge about total laryngectomy | 30 days after hospital discharge (approximately 7 weeks after registration)
  -The change in knowledge due to the educational intervention will be measured using a within subject comparison of patient pre- and post-education test scores (e.g. each patient's post-education scores minus preeducation scores).

CONTACTS AND LOCATIONS:
Overall Officials: Brian Nussenbaum, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu